CLINICAL TRIAL: NCT01687764
Title: Combination of Active or Placebo Attentional Bias Modification Treatment (ABMT) to Either Cognitive Behavioral Group Therapy (CBGT) or Psychoeducational Control Intervention (PCI) for Anxiety Disorders in Children: a Randomized Clinical Trial
Brief Title: Combination of Active or Placebo Attentional Bias Modification Treatment (ABMT) to Either Cognitive Behavioral Group Therapy (CBGT) or Psychoeducational Control Intervention (PCI) for Anxiety Disorders in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCPA11-0249
Record Dates: First submitted 2011-10-26; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Generalized Anxiety Disorder; Separation Anxiety Disorder; Social Anxiety Disorder
Keywords: Generalized Anxiety Disorder (GAD); Separation Anxiety Disorder (SeAD); Social Anxiety Disorder (SoAD)
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Social | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- CBGT+ABMT(active) (Experimental)
  Interventions: Other: Attentional Bias Modification Treatment (ABMT) - Active; Behavioral: Cognitive Behavioral Group Therapy
- CBGT+ABMT(placebo) (Experimental)
  Interventions: Other: Attentional Bias Modification Treatment - Placebo; Behavioral: Cognitive Behavioral Group Therapy
- PCI+ABMT(active) (Experimental)
  Interventions: Other: Attentional Bias Modification Treatment (ABMT) - Active; Behavioral: Psychoeducational Control Intervention
- PCI+ABMT(placebo) (Placebo Comparator)
  Interventions: Other: Attentional Bias Modification Treatment - Placebo; Behavioral: Psychoeducational Control Intervention

INTERVENTIONS:
Other: Attentional Bias Modification Treatment (ABMT) - Active — The ABMT consists of 160 trials (120 angry-neutral and 40 neutral-neutral presentations). In the ABM condition, the target appears at the neutral-face location in all angry-neutral trials. Probe type (< or >) is not factorially counterbalanced but appears with equal probability for each of the following: angry-face location, probe location, or actor.
  Arms: CBGT+ABMT(active); PCI+ABMT(active)
Other: Attentional Bias Modification Treatment - Placebo — The Placebo protocol consists of 160 trials (120 angry-neutral and 40 neutral-neutral presentations). In the placebo condition, angry-face location, probe location, and actor are fully counterbalanced in presentation.
  Arms: CBGT+ABMT(placebo); PCI+ABMT(placebo)
Behavioral: Cognitive Behavioral Group Therapy — "FRIENDS for Life" Australian protocol for the treatment of anxiety disorders in children
  Arms: CBGT+ABMT(active); CBGT+ABMT(placebo)
Behavioral: Psychoeducational Control Intervention — Psychoeducational control intervention provides only brief psychoeducational information about anxiety associated with general educational activities
  Arms: PCI+ABMT(active); PCI+ABMT(placebo)

SUMMARY:
The objective of this project is to test the combination of active or placebo Attentional Bias Modification Treatment (ABMT) to either Cognitive Behavioral Group Therapy (CBGT) or Psychoeducational Control Intervention (PCI) for anxiety disorders in children.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Generalized Anxiety Disorder (GAD), Separation Anxiety Disorder (SeAD) or Social Anxiety Disorder (SoAD) according to KSADS-PL psychiatric interview

Exclusion Criteria:

* Other psychiatric disorder that causes more impairment and suffering than GAD, SeAD or SoAD in the clinical evaluation
* Current or previous treatment (behavioral or pharmacological) for a psychaitric disorder in childhood
* IQ < 70 (Raven)

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) / continuous | Endpoint (week 10) and 6-month follow-up
  Score change on Pediatric Anxiety Rating Scale (PARS) from baseline to week 10 and to 6-month follow-up
Clinical Global Impression - Improvement Scale (CGI-I) / dichotomous | Endpoint (week-10) and 6-month follow-up
  Percentage of subjects with less than 2 points in the CGI-I scale in week 10 and in 6-month follow-up

SECONDARY OUTCOMES:
Screen for Children and Anxiety Related Emotional Disorders (SCARED) | Endpoint (week-10) and 6-months follow-up
  Score change in SCARED child and parent versions from baseline to week 10 and 6-months follow-up
Childhood Depression Inventory (CDI) | Endpoint (week-10) and 6-month follow-up
  Score change in CDI from baseline to week-10 and to 6-month follow-up
Swanson, Nolan, and Pelham scale - Version IV (SNAP-IV) | Endpoint (week-10) and 6-month follow-up
  Score change in SNAP-IV from baseline to week-10 and 6-month follow-up
Spence Children's Anxiety Scale (SCAS) | Endpoint (week-10) and 6-month follow-up
  Score change in SCAS from baseline to week-10 and to 6-month follow-up
Neuropsychological measures | Endpoint (week-10) and 6-month follow-up
  Change in neuropsychological measures from baseline to week-10 and 6-month follow-up
Biological measures | Endpoint (week-10) and 6-month follow-up
  Change in biological measures from baseline to week-10 and to 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gisele G Manfro, MD, PhD, Principal Investigator — Federal University of Rio Grande do Sul / Hospital de Clínicas de Porto Alegre; Silvia H Koller, PhD, Principal Investigator — Federal University of Rio Grande do Sul / University of Psychology
Locations (4):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States
- University of Queensland, Brisbane Saint Lucia, Queensland, Australia
- Federal University of Rio Grande do Sul / Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil
- Tel-Aviv University, Tel Aviv, Israel